CLINICAL TRIAL: NCT01907646
Title: Role of Bladder Training During Post-operative Hospital Stay After Radical Hysterectomy in Patients: a Randomized Trial
Brief Title: Role of Bladder Training During Post-operative Hospital Stay After Radical Hysterectomy in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2012-08-18; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Uterine Cervical Neoplasms
Keywords: bladder training, radical hysterectomy,gynaecologic cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bladder training group (Experimental): The patients of this group were submitted to passive vesical gymnastic during the second and third postoperative days, throughout the closure of the catheter for 3 h and open it for 15 min all day long.
  Interventions: Device: bladder training
- No bladder training group (Experimental): The patients of this group were not submitted to passive vesical gymnastic during the second and third postoperative days
  Interventions: Procedure: No bladder training

INTERVENTIONS:
Device: bladder training — vescical catheter
  Arms: Bladder training group
Procedure: No bladder training
  Arms: No bladder training group

SUMMARY:
The objective of the study is to evaluate the impact and the outcome of bladder training during post-operative hospital stay after radical hysterectomy, mainly after neoadjuvant concurrent chemo-radiation therapy for locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

- Women who underwent Querleu-Morrow class B2 and class C1 RH were enrolled in this randomized prospective study.

Exclusion Criteria:

-All the patients with preoperative urinary dysfunctions were excluded by study. Other exclusion criteria were surgery of lower urinary tract and psychiatric disease.

Ages: 27 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
clean intermittent self-catheterization | three days
  necessity and duration of clean intermittent self-catheterization after three days

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy, Italy